CLINICAL TRIAL: NCT06809582
Title: Does the Positioning in Retrograde Intrarenal Surgery Affect Stone-Free Rates? A Prospective Randomized Controlled Trial
Brief Title: Impact of Surgical Position on Stone-Free Rates in Retrograde Intrarenal Surgery
Acronym: POS-RIRS-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Murat Gulsen, Assistant professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B.30.2.ODM.0.20.08/603-670
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Stone, Kidney; Stones, Kidney; Stone;Renal
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard lithotomy position (No Intervention): In this arm we will use standard lithotomy position as control group.
- T-Tilt Lithotomy Position (Active Comparator)
  Interventions: Procedure: The T-Tilt position

INTERVENTIONS:
Procedure: The T-Tilt position — The T-Tilt position is a modified lithotomy position used during retrograde intrarenal surgery (RIRS). In this position:
  The patient is placed in a 30-degree Trendelenburg position, meaning the head is slightly lower than the feet.
  The surgical side is elevated at a 30-degree angle to improve access to the kidney.
  This modified positioning is designed to enhance stone clearance, particularly by facilitating the movement of stone fragments away from the lower kidney calyces, where residual stones often remain. Researchers will compare this position to the standard lithotomy position to determine its impact on stone-free rates and surgical outcomes.
  Arms: T-Tilt Lithotomy Position

SUMMARY:
The goal of this clinical trial is to determine whether the surgical position during retrograde intrarenal surgery (RIRS) affects stone-free rates in adults with kidney stones. The main questions it aims to answer are:

* Does the modified lithotomy position result in a higher stone-free rate compared to the standard lithotomy position?
* Are there differences in complication rates between the two surgical positions?

Researchers will compare patients undergoing RIRS in the standard lithotomy position to those in the modified lithotomy position (30-degree Trendelenburg with elevated surgical side) to assess its impact on stone clearance and surgical outcomes.

Participants will:

* Be randomly assigned to one of two surgical positions
* Undergo RIRS with standard surgical procedures
* Have follow-up imaging to assess stone clearance after surgery

This study aims to improve surgical techniques and patient outcomes in kidney stone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of single or multiple kidney stones, with the largest stone ≤2 cm
* Age ≥18 years
* Provided written informed consent to participate in the study
* Indicated for retrograde intrarenal surgery (RIRS) as a treatment approach

Exclusion Criteria:

* Severe cardiovascular disease (e.g., heart failure)
* Congenital kidney anomalies (e.g., horseshoe kidney, ectopic kidney)
* Concurrent ureteral stones
* Pregnancy or planning pregnancy
* History of previous kidney surgery on the same side
* Active urinary tract infection (UTI)
* Coagulopathy or use of anticoagulant therapy that cannot be stopped before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Stone-Free Rate After Retrograde Intrarenal Surgery | 6 weeks post-surgery
  The percentage of participants with no residual kidney stones (≤4 mm fragments) on non-contrast computed tomography (CT) at 6 weeks postoperatively.

SECONDARY OUTCOMES:
Postoperative Complication Rate | Within 30 days post-surgery
  he percentage of participants experiencing any postoperative complications, classified according to the Clavien-Dindo grading system.

OTHER OUTCOMES:
Rehospitalization Rate | Within 30 days post-surgery
  The percentage of participants requiring hospital readmission due to complications related to the surgical procedure
Total Laser Energy Used | Intraoperative
  The total Holmium:YAG laser energy (Joules) applied during stone fragmentation

CONTACTS AND LOCATIONS:
Overall Officials: Murat Gulsen, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Canakci C, Dincer E, Can U, Coskun A, Otbasan BK, Ozkaptan O. The relationship between stone-free and patient position in retrograde intrarenal surgery: a randomized prospective study. World J Urol. 2024 May 9;42(1):308. doi: 10.1007/s00345-024-05013-1. PMID 38722376
- [Result] Liaw CW, Khusid JA, Gallante B, Bamberger JN, Atallah WM, Gupta M. The T-Tilt Position: A Novel Modified Patient Position to Improve Stone-Free Rates in Retrograde Intrarenal Surgery. J Urol. 2021 Nov;206(5):1232-1239. doi: 10.1097/JU.0000000000001948. Epub 2021 Jul 12. PMID 34251886

DOCUMENTS (2):
  • Statistical Analysis Plan (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT06809582/SAP_000.pdf
  • Informed Consent Form (2024-11-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT06809582/ICF_001.pdf